CLINICAL TRIAL: NCT00082407
Title: Efficacy of Exenatide (AC2993, Synthetic Exendin-4, LY2148568) Compared With Twice-Daily Biphasic Insulin Aspart in Patients With Type 2 Diabetes Using Sulfonylurea and Metformin
Brief Title: Exenatide Compared With Twice-Daily Biphasic Insulin Aspart in Patients With Type 2 Diabetes Using Sulfonylurea and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWAD
Record Dates: First submitted 2004-05-06; First posted 2004-05-10 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; exendin; Amylin; Lilly; insulin aspart
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Arm (Experimental): subcutaneous injection, twice daily; 5 mcg for 4 weeks followed by 10 mcg for 48 weeks
  Interventions: Drug: exenatide
- Biphasic Insulin Aspart Arm (Active Comparator): subcutaneous injection, twice daily; titration to target blood glucose level
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, twice daily; 5 mcg for 4 weeks followed by 10 mcg for 48 weeks
  Other Names: Byetta
  Arms: Exenatide Arm
Drug: biphasic insulin aspart — subcutaneous injection, twice daily; titration to target blood glucose level
  Other Names: NovoLog
  Arms: Biphasic Insulin Aspart Arm

SUMMARY:
This is a Phase 3, multicenter, open-label, comparator-controlled trial comparing the effect of exenatide twice daily to twice daily biphasic insulin aspart on glycemic control, as measured by hemoglobin A1c (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Patients have been treated with a stable dose of the following for at least 3 months prior to screening: 1. >=1500 mg/day immediate-release metformin or extended-release metformin and at least an optimally effective dose for brand of sulfonylurea, or 2. a fixed-dose sulfonylurea/metformin combination therapy with the same sulfonylurea and metformin requirements as for the individual components
* HbA1c between 7.0% and 11.0%, inclusive.
* Patients have a body mass index >25kg/m2 and <40 kg/m2.
* Female patients are not breastfeeding, and female patients of childbearing potential test negative for pregnancy, do not intend to become pregnant during the study, and agree to continue using a reliable method of birth control

Exclusion Criteria:

* Patients are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study.
* Patients are employed by Lilly or Amylin.
* Patients have previously, in this or any other study, received exenatide or glucagon-like peptide-1 analogs.
* Patients have participated in an interventional medical, surgical, or pharmaceutical study within 30 days prior to screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.
* Patients have had greater than three episodes of severe hypoglycemia within 6 months prior to screening.
* Patients have less than 5 years of remission history from any malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer).
* Patients have cardiac disease that is Class III or IV, according to the New York Heart Association criteria.
* Patients have a known allergy or hypersensitivity to biphasic insulin aspart, exenatide, or excipients contained in these agents.
* Patients have characteristics contraindicating metformin or sulfonylurea use, according to product-specific label.
* Patients have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine >=1.5 mg/dL for males and >=1.2 mg/dL for females.
* Patients have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine aminotransferase/serum glutamic pyruvic transaminase greater than three times the upper limit of the reference range.
* Patients have known hemoglobinopathy or chronic anemia.
* Patients have active proliferative retinopathy or macular edema.
* Patients are receiving treatment for gastrointestinal disease with a drug directly affecting gastrointestinal motility, including but not limited to metoclopramide, cisapride, and chronic macrolide antibiotics.
* Patients are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to screening.
* Patients have used any prescription drug to promote weight loss within 3 months prior to screening.
* Patients have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to screening: insulin, thiazolidinediones, alpha-glucosidase inhibitors, meglitinides.
* Patients have any other condition (including known drug or alcohol abuse or psychiatric disorder) that precludes them from following and completing the protocol, in the opinion of the investigator.
* Patients fail to satisfy the investigator of suitability to participate for any other reason.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2003-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (69):
- Croatia (4):
  - Clinical Hospital Osijek, Osijek
  - Klinica bolnica Dubrava, Zagreb
  - Klinicki bolnicki centar Zagreb-Rebro, Zagreb
  - Opca bolnica "Sveti Duh", Zagreb
- Germany (13):
  - Internistische Gemeinschaftspraxis, Augsburg
  - Dr. Karlheinz Hehemann, Beckum
  - Dr. Klaus Busch, Dortmund
  - Medical Clinic and Policlinic 3, Giessen
  - Diabetologische Schwerpunktpraxis, Hamburg
  - IKFE GmbH, Mainz
  - Institut for diabetic research, Munich
  - Profil, Institut fur Stoffwechselstorungen, Neuss
  - Dr. Thomas Behnke, Neuwied
  - Dr. Bernd Donaubauer, Oschatz
  - Marienhospital Osnabruck, Osnabrück
  - Dr. Joerg Steindorf, Schkeuditz
  - Dr. Jerzi Jasinski, Wiesbaden
- Greece (5):
  - "Polyclinic" General Hospital of Athens, Athens
  - Department of Endocrinology, Athens
  - Diabetes Center, Athens
  - University Hospital of Patras, Pátrai
  - 1st Internal Medicine Department "Papagergiou", Thessaloniki
- Italy (6):
  - Instituto di Endocrinologia, Catania
  - Dipartimento di fisiopatologia clinica, Florence
  - U.O. Medicina Generale, Milan
  - Ospedale Civile di Padova, Padua
  - Policlinico Univarsitario P. Giaccone, Palermo
  - U.O. Universita di Malattie del Metabolismo e Diabetologia, Torino
- Netherlands (3):
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Maxima Medisch Centrum Location Eindhoven, Eindhoven
- Portugal (4):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Santo Andre, Leiria
  - Associacao Protectora dos Diabeticos de Portugal, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
- Romania (3):
  - Spitalul Judetean Brasov, Brasov
  - Institutul de Diabet, Bucharest
  - Spitalul Clinic nr. 1 Judetean, Judet Timis
- Russia (7):
  - National Endocrinology Research Center, Moscow
  - Setchenov Moscow Medical Academy, Moscow
  - Moscow State Medical Stomatological, Moscow
  - Russian Medical Academy for Advanced Medical Studies, Ministry of Health, Moscow
  - Hospital of St. Elizabeth's, Saint Petersburg
  - City Clinical Hospital #2, Saint Petersburg
  - Medical Military Academy, Saint Petersburg
- Slovenia (2):
  - Univerzitetni klinicni center Ljubljana, Ljubljana
  - Splosna bolnisnica Maribor, Maribor
- Spain (6):
  - Hospital Vega Baja, Alicante
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Endocrinology Service (Planta Baja), Palma de Mallorca
  - Hospital Virgen de Valme, Seville
  - Hospital General de Teruel, Teruel
  - Hospital la Ribera Alzira, Valencia
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Tzu Chi General Hospital, Hualien City
  - Veteran General Hospital-Taichung, Taichung
  - Tri-Service General Hospital, Taipei
- United Kingdom (12):
  - Diabetes Research, Ward 34, Birmingham Heartlands Hospital, Birmingham
  - Diabetes Unit, Blackburn Royal Infirmary, Blackburn
  - Colchester General Hospital, Colchester
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - The Michael White Center for Diabetes and Endocrinology, Hull
  - Clinical Sciences Centre, Liverpool
  - Education Centre, James Cook University Hospital, Middlesbrough
  - Wellcome Labs, Royal Victoria Infirmary, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham
  - Diabetes Trial Unit OCDEM, Churchill Hospital, Oxford
  - Diabetes Unit, Gladsone Centre, Maelor Hospital, Wrexham

REFERENCES:
- [Result] Nauck MA, Duran S, Kim D, Johns D, Northrup J, Festa A, Brodows R, Trautmann M. A comparison of twice-daily exenatide and biphasic insulin aspart in patients with type 2 diabetes who were suboptimally controlled with sulfonylurea and metformin: a non-inferiority study. Diabetologia. 2007 Feb;50(2):259-67. doi: 10.1007/s00125-006-0510-2. Epub 2006 Dec 8. PMID 17160407
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four patients withdrew from the study prior to receiving study drug.
Period: Overall Study
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Started | 255 | 250
Received Treatment (Intent to Treat) | 253 | 248
Completed | 199 | 223
Not Completed | 56 | 27
Not completed — Adverse Event | 20 | 0
Not completed — Protocol Violation | 14 | 12
Not completed — Patient Decision | 13 | 6
Not completed — Physician Decision | 5 | 3
Not completed — Loss of Glucose Control | 2 | 2
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: IIT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm | Total
Number analyzed (Participants) | 253 | 248 | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 174 | 358
  >=65 years | 69 | 74 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.7) | 58.5 (9.2) | 58.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 122 | 257
  Male | 118 | 126 | 244

OUTCOME MEASURES:

1. Primary Outcome: Change in Glcosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline to week 52
Time Frame: baseline, week 52
Population: Last Observation Carried Forward; Intent to Treat, computed from the patients having both baseline and post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 248 | 246
percentage
  Baseline HbA1c | 8.59 (0.07) | 8.65 (0.07)
  Change in HbA1c at week 52 | -0.98 (0.07) | -0.88 (0.07)
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Non-Inferiority or Equivalence — Pre-specified non-inferiority margin was 0.4% (i.e., noninferiority is demonstrated if the upper limit of a two-sided 95% confidence interval for the difference in change in HbA1c between exenatide and biphasic insulin aspart is less than 0.4%.); p = 0.2534, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI [-0.28 to 0.08]

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7%
Description: Percentage of patients in each arm who had HbA1c >7% at baseline and had HbA1c <=7% at week 52 (percentage = [number of subjects with HbA1c <=7% at week 52 divided by number of subjects with HbA1c >7% at baseline] * 100%).
Time Frame: 52 weeks
Population: Last Observation Carried Forward; Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 227 | 237
percentage of participants | 31.7 | 24.1
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Superiority or Other; p = 0.0779, Fisher Exact

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 52.
Time Frame: baseline, week 52
Population: Intent to Treat, computed from the patients having both baseline and week 52 data.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 205 | 223
kg
  Baseline body weight | 85.51 (0.99) | 83.38 (0.99)
  Change in body weight at week 52 | -2.54 (0.17) | 2.92 (0.17)
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Superiority or Other; p = 0.0001, ANCOVA

4. Secondary Outcome: Change in Fasting Serum Glucose
Description: Change in fasting serum glucose from baseline to week 52
Time Frame: baseline, week 52
Population: Intent to Treat, computed from the patients having both baseline and week 52 data.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 198 | 218
mmol/L
  Baseline fasting serum glucose | 11.00 (0.18) | 11.30 (0.18)
  Change in fasting serum glucose at week 52 | -1.75 (0.19) | -1.64 (0.19)
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Superiority or Other; p = 0.6456, ANCOVA

5. Secondary Outcome: Change in 7-point Self-monitored Blood Glucose (SMBG) Profile
Description: Change in 7-point (pre-breakfast, after breakfast, pre-lunch, after lunch, pre-dinner, after dinner, 0300 hours) SMBG profile from baseline to week 52
Time Frame: baseline, week 52
Population: Last Observation Carried Forward; Intent to Treat
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 253 | 248
mmol/L
  Pre-breakfast: Baseline SMBG | 9.57 (2.34) | 9.86 (2.65)
  Pre-breakfast: Change in SMBG at week 52 | -1.15 (2.60) | -1.68 (2.33)
  After breakfast: Baseline SMBG | 12.30 (3.02) | 12.71 (3.03)
  After breakfast: Change in SMBG at week 52 | -3.83 (3.30) | -3.06 (3.26)
  Pre-lunch: Baseline SMBG | 9.38 (2.86) | 9.86 (3.30)
  Pre-lunch: Change in SMBG at week 52 | -1.47 (3.01) | -2.40 (3.44)
  After lunch: Baseline SMBG | 11.18 (3.14) | 11.39 (3.58)
  After lunch: Change in SMBG at week 52 | -1.72 (3.48) | -1.76 (3.74)
  Pre-dinner: Baseline SMBG | 9.35 (2.86) | 9.57 (3.03)
  Pre-dinner: Change in SMBG at week 52 | -1.06 (3.25) | -1.52 (3.42)
  After dinner: Baseline SMBG | 11.25 (3.04) | 11.68 (3.27)
  After dinner: Change in SMBG at week 52 | -3.11 (3.76) | -2.44 (3.69)
  3:00 AM: Baseline SMBG | 9.08 (2.63) | 9.58 (3.14)
  3:00 AM: Change in SMBG at week 52 | -0.96 (3.14) | -1.95 (3.13)

6. Secondary Outcome: Percentage of Patients With Hypoglycemic Events
Description: Percentage of patients who experienced at least one episode of hypoglycemia at any point during the 52 week Parent Study (incidence of hypoglycemia = number of patients who experienced at least one episode of hypoglycemia at any point during the 52 week Parent Study divided by the total number of patients who particiapted in the 52 week Parent Study
Time Frame: 52 weeks
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 253 | 248
percentage of participants | 53.0 | 51.6
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Superiority or Other; p = 0.7888, Fisher Exact

7. Secondary Outcome: Change in Rate of Hypoglycemic Events
Description: Change in rate of hypoglycemic events per 30 days per patient from baseline to week 52
Time Frame: baseline, week 52
Population: Last Observation Carried Forward; Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: events per 30 days per patient
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Number analyzed (Participants) | 253 | 248
events per 30 days per patient
  Baseline event rate | 0.22 (0.07) | 0.18 (0.07)
  Change in event rate at week 52 | 0.19 (0.06) | 0.26 (0.06)
Statistical Analysis 1: Comparison: Exenatide Arm vs Biphasic Insulin Aspart Arm; Test type: Superiority or Other; p = 0.3722, ANCOVA

ADVERSE EVENTS:
Arm/Group | Exenatide Arm | Biphasic Insulin Aspart Arm
Serious Adverse Events (participants affected / at risk) | 19 | 11
Other Adverse Events (participants affected / at risk) | 179 | 128
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exenatide Arm | Biphasic Insulin Aspart Arm
Anemia (Blood and lymphatic system disorders) | 2/253 | 0/248
Angina pectoris (Cardiac disorders) | 2/253 | 0/248
Myocardial infarction (Cardiac disorders) | 2/253 | 0/248
Atrial fibrillation (Cardiac disorders) | 1/253 | 0/248
Coronary artery disease (Cardiac disorders) | 1/253 | 0/248
Acute coronary syndrome (Cardiac disorders) | 0/253 | 1/248
Atrial flutter (Cardiac disorders) | 0/253 | 1/248
Bundle branch block left (Cardiac disorders) | 0/253 | 1/248
Vertigo (Ear and labyrinth disorders) | 0/253 | 1/248
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1/253 | 0/248
Nausea (Gastrointestinal disorders) | 1/253 | 0/248
Anal fistula (Gastrointestinal disorders) | 0/253 | 1/248
Asthenia (General disorders) | 1/253 | 0/248
Calcinosis (General disorders) | 1/253 | 0/248
Gait disturbance (General disorders) | 1/253 | 0/248
Abdominal wall abscess (Infections and infestations) | 1/253 | 0/248
Appendicitis (Infections and infestations) | 1/253 | 0/248
Cellulitus (Infections and infestations) | 1/253 | 0/248
Injection site cellulitus (Infections and infestations) | 1/253 | 0/248
Lobar pneumonia (Infections and infestations) | 0/253 | 1/248
Fall (Injury, poisoning and procedural complications) | 1/253 | 0/248
Radius fracture (Injury, poisoning and procedural complications) | 1/253 | 0/248
Weight decreased (Investigations) | 1/253 | 0/248
Anorexia (Metabolism and nutrition disorders) | 1/253 | 0/248
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/253 | 0/248
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/253 | 0/248
Neck pain (Musculoskeletal and connective tissue disorders) | 0/253 | 1/248
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/253 | 1/248
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/253 | 1/248
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/253 | 1/248
Cognitive disorder (Nervous system disorders) | 1/253 | 0/248
Cerebrovascular accident (Nervous system disorders) | 0/253 | 1/248
Major depression (Psychiatric disorders) | 1/253 | 0/248
Urinary incontinence (Renal and urinary disorders) | 0/253 | 1/248
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/253 | 0/248
Breast microcalcification (Reproductive system and breast disorders) | 0/253 | 1/248
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1/253 | 0/248
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0/253 | 1/248
Hematoma (Vascular disorders) | 1/253 | 0/248
Hypertension (Vascular disorders) | 1/253 | 0/248
Peripheral ischemia (Vascular disorders) | 1/253 | 0/248
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide Arm | Biphasic Insulin Aspart Arm
Nausea (Gastrointestinal disorders) | 84/253 | 1/248
Vomiting (Gastrointestinal disorders) | 38/253 | 8/248
Nasopharyngitis (Infections and infestations) | 28/253 | 24/248
Diarrhea (Gastrointestinal disorders) | 24/253 | 5/248
Influenza (Infections and infestations) | 18/253 | 16/248
Headache (Nervous system disorders) | 12/253 | 13/248
Hypoglycemia (Metabolism and nutrition disorders) | 134/253 | 128/248

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days